CLINICAL TRIAL: NCT06510699
Title: Randomized Clinical Trial to Evaluate the Use of Genotype-based Dosing of Voriconazole in Patients With Haematological Malignancy
Brief Title: Pharmacogenomics for Better Treatment of Fungal Infections in Cancer
Acronym: PRAGMATIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Metro North Hospital and Health Service (Unknown); Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other); University of Sydney (Other); Western Sydney Local Health District (Other); Sydney Children's Hospitals Network (Other); Peter MacCallum Cancer Centre, Australia (Other); University of Melbourne (Other); Royal Adelaide Hospital (Other); Pathology Queensland (Unknown); Royal Brisbane and Women's Hospital (Other Government); Lady Cilento Children's Hospital, Brisbane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAGMATIC 01
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Fungal Infection; Haematological Malignancy; Blood Cancer; Infectious Disease
Keywords: infection; cancer; pharmacogenomic; genotype-based dosing; CYP2C19
MeSH Terms: conditions — Mycoses; Hematologic Neoplasms; Communicable Diseases; Infections; Neoplasms

STUDY DESIGN:
Intervention Model Description: PRAGMATIC is a parallel-group randomised (1:1) clinical trial aiming to recruit at least 104 patients. A hybrid feasibility sub-study will assess the scalability of genotype directed dosing to ensure a sustainable integration of the interventions into the clinical workflow. A health economic sub-study will evaluate the costs, health outcomes and cost effectiveness of genotype-directed testing compared to standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Precision Care (Experimental): Voriconazole dosing will be initiated using current standard care dosing. Samples for TDM and genotype testing will be collected. Based on the results of these tests on Day 5, 8, 14, and up to day 30 ( ± 1 day) patients will be evaluated for dose adjustment using dosing software that includes patient data including TDM and genotype data.
  Interventions: Other: genotype-directed dosing with dosing software based on therapeutic drug monitoring
- Standard Care (No Intervention): Current standard of care at trial-site institutions uses weight-based (mg/kg) initial dosing of voriconazole, with dose adjustment based on standard therapeutic drug monitoring (TDM) results of measured voriconazole concentrations and based on clinical judgement.

INTERVENTIONS:
Other: genotype-directed dosing with dosing software based on therapeutic drug monitoring — Genotype-directed dosing with dosing software based on therapeutic drug monitoring
  Other Names: genotype directed with dosing software
  Arms: Precision Care

SUMMARY:
This project aims to address invasive fungal infections in patients with blood cancer, by precision dosing of voriconazole based on CYP2C19 genotype testing with Bayesian dose-forecasting dosing software to develop patient-centric and maximally effective dosing regimens. This study investigates if voriconazole increases the proportion of patients achieving therapeutic exposure at day 8 of dosing compared with standard care; and will assess factors that influence the implementation of genotype testing and dosing software in the healthcare system, including fidelity, feasibility, acceptability and cost-effectiveness. It will recruit at least 104 kids and adults in a parallel-group randomised clinical trial. A hybrid feasibility sub-study will assess the scalability of genotype-directed dosing to ensure sustainable integration of the interventions into the clinical workflow. A health economic sub-study will evaluate the costs, health outcomes and cost-effectiveness of genotype-directed testing compared to standard care.

DETAILED DESCRIPTION:
Participants will be randomly assigned to standard care or precision care. Current standard of care at trial-site institutions uses weight-based (mg/kg) initial dosing of voriconazole, with dose adjustment based on standard therapeutic drug monitoring (TDM) results of measured voriconazole concentrations based on clinical judgement. In precision care, voriconazole dosing will be initiated using current standard dosing. Samples for the TDM and genotype testing will be collected. Based on results of these tests on Day 5 (+/- 1 day) patients will be evaluated for dose adjustment using dosing software that includes patient data, TDM and genotype data.

Trial procedures: following baseline data collection and randomisation genotype testing will be performed on Day 1. The precision care group have dose adjustment performed on Days 5, 9, 15, and 22 using genotype and/or TDM results in dosing software. The standard care group will have TDM performed, and dose adjustments in accordance with usual clinical practice. Blood sampling for TDM will be performed 24-hours prior to dose adjustment, with additional blood samples collected on Days 1 and 2 in both standard care and precision care groups. All blood sampling, genotype testing and dose adjustments will be performed +/- day to support feasibility.

The primary objective is to compare the proportion of patients achieving therapeutic voriconazole exposure at Day 8 when using precision care compared to standard care.

Secondary objectives are:

1. Clinical: comparison of clinical success of voriconazole treatment between precision care and standard care groups, where clinical success is defined as an absence of clinical deterioration or event that requires a change of therapy.
2. Antifungal exposure: to compare antifungal exposure over the first 28 days of therapy between precision care and standard care groups.
3. Comparative precision care methodologies: compare if there is a difference in daily dose recommendations between using a genotype nomogram, dosing software with TDM, or a combination of dose adjustment in precision care.
4. Feasibility of precision care interventions: to determine if it is feasible to perform the measurement of voriconazole concentrations and genotype testing for use in dosing software in time to intervene prior to Day 5 and/or Day 9 dose adjustment.
5. Genotype: describe clinical success of voriconazole between genotypes.

The implementation feasibility sub-study will assess the scalability of precision care to support optimal voriconazole dosing by tailoring the intervention to each trial setting and measuring outcomes with the involvement of key stakeholders (end-users, health administrators, consumers, community members).

Data will be collected to ascertain Fidelity including: 1) assess barriers and enablers; 2) identify prioritise the factors influencing delivery and tailor these to fit local settings; 3) assess intended fidelity to the precision care intervention.

Data will be collected to ascertain Feasibility or the extent to which precision care can be successfully used in each study setting via completion of the feasibility implementation measure (FIM) at baselines and quarterly thereafter, including qualitative interviews at the end of the study.

Data will be collected to ascertain Acceptability or whether end-users perceive precision care as agreeable or satisfactory by survey and qualitative interviews with pharmacists, physicians and health administrators.

Data will be collected to undertake an economic evaluation to determine the cost-effectiveness of precision versus standard care, exploring individual level data, incremental cost effectiveness ratios (ICERs) at day 14 and 30; and cost-utility analysis to demonstrate if precision care offers value for money at Day 30 in the Australian setting. The health economic evaluation will include use of surveys to capture: 1) healthcare usage of trial participants; 2) implementation feasibility measures; and 3) implementation costs.

Data will be collected to ascertain scalability or the ability to expand the efficacy of precision care on a small scale in controlled conditions to real world conditions to a greater proportion of the population.

Therapeutic trough voriconazole exposures (concentrations) In this trial, serum concentrations > 1 mg/L (minimum effective concentration) and < 5 mg/L (maximum safe concentration) are defined as the therapeutic range. Treating clinicians may nominate an individualised patient target within this range prior to randomisation and that range will be applied during the trial. Where dosing software is being applied, the software will be programmed to target 2.5 mg/L.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years.
* Written informed consent obtained.
* Decision to prescribe voriconazole.
* Diagnosed with haematological malignancy or disorder.
* Admitted to a trial site, or sufficient outpatient follow-up appointments are feasible

Exclusion Criteria:

* Post-allogeneic haematopoietic stem cell transplant (HCT) patient, without access to pre HCT DNA
* Death is likely imminent within 7 days.
* Previously randomised to this trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Therapeutic trough voriconazole concentration at Day 8 | Day 8
  Proportion of patients with measured therapeutic trough voriconazole concentration at Day 9 (+/- 1 day)

SECONDARY OUTCOMES:
Simulated therapeutic trough voriconazole exposure at Day 8 | Day 8
  Proportion of patients with simulated therapeutic trough voriconazole exposure at Day 8
Measured therapeutic trough voriconazole exposure at Day 14. | Day 14
  Proportion of patients with measured therapeutic trough voriconazole exposure at Day 14.
Simulated therapeutic trough voriconazole exposure at Day 14 | Day 14
  Proportion of patients with simulated therapeutic trough voriconazole exposure at Day 14
Measured therapeutic trough voriconazole exposure at both Days 8 and 14 | Days 8 and 14
  Proportion of patients with measured therapeutic trough voriconazole exposure at both Days 8 and 14
Simulated therapeutic trough voriconazole exposure at both Days 8 and 14 | Days 8 and 14
  Proportion of patients with simulated therapeutic trough voriconazole exposure at both Days 8 and 14
Simulated therapeutic trough voriconazole exposure from Day 8 to Day 30 | Day 8 to Day 30
  Proportion of patients with simulated therapeutic trough voriconazole exposure from Day 8 to Day 30
Days to achieve first measured therapeutic trough voriconazole exposure | Assessed over 30 days
  Number of days to achieve first measured therapeutic trough voriconazole exposure
Doses to achieve first measured therapeutic trough voriconazole exposure. | Assessed over 30 days
  Number of doses to achieve first measured therapeutic trough voriconazole exposure.
Percent difference in dose when dose adjustment is performed | Assessed over 30 days
  Percent difference in dose when dose adjustment is performed (i) on the first occasion and (ii) on subsequent occasions (set to 0 if no adjustment).
Number of days of antifungal therapy | Assessed over 30 days
  Number of days of antifungal therapy
Number of doses of antifungal therapy | Assessed over 30 days
  Number of doses of antifungal therapy
Clinical cure or stable disease | Assessed over 30 days
  Proportion of patients achieving invasive fungal disease (IFD) clinical cure or stable disease; defined by treating team, if indication is IFD treatment
Patients with no reported fungal infection during course | Assessed over 30 days
  Proportion of patients with no reported fungal infection during course, if indication is IFD prophylaxis.
Hospital free days | Day 30
  Number of hospital free days at day 30
Length of hospital stay post-randomisation | Assessed over 30 days
  Length of hospital stay post-randomisation
Number of patients experiencing at least one adverse event | Assessed over 30 days
  Number of patients experiencing at least one adverse event
Number and type of adverse events | Assessed over 30 days
  Number and type of adverse events
All-cause mortality at 30 days | Assessed over 30 days
  All-cause mortality at 30 days
Clinical success | Assessed over 30 days
  Proportion of patients achieving clinical success, defined as an absence of a clinical deterioration or event that requires a change of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, PhD, Principal Investigator — The University of Queensland
Locations (7):
- Fred Hutchinson Cancer Centre, Seattle, Washington, United States
- Australia (6):
  - Sydney Children's Hospital Network, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Children's Hospital Queensland, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided